CLINICAL TRIAL: NCT04598230
Title: Partners in Caring for Anxious Youth
Acronym: PCAY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Cincinnati (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John T Walkup, MD, Department Chair Pritzker Department of Psychiatry, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20203537
Record Dates: First submitted 2020-09-23; First posted 2020-10-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Anxiety, Separation; Anxiety, Generalized; Anxiety, Social
Keywords: anxiety disorders; child; adolescent; pediatric; cognitive behavioral therapy; selective serotonin reuptake inhibitor; antidepressant medication
MeSH Terms: conditions — Anxiety, Separation; Generalized Anxiety Disorder; Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Psychotherapy; Combined Modality Therapy; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination therapy (COMB) (Active Comparator): Participants randomized to this arm will receive cognitive behavioral therapy and one of three study medications (fluoxetine, sertraline, or escitalopram).
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Drug: Combination therapy (COMB)
- Cognitive behavioral therapy (CBT) (Active Comparator): Participants randomized to this arm will receive cognitive behavioral therapy (CBT) only
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants randomized to this arm will receive up to 20 sessions of evidence based cognitive behavioral therapy (CBT) of extended duration, with more exposure tasks and greater family involvement than has been studied in the past.
  Other Names: CBT; psychotherapy
Drug: Combination therapy (COMB) — Participants randomized to this arm will receive cognitive behavioral therapy comparable to that in the cognitive behavioral therapy arm, plus one of three selective serotonin reuptake inhibitors (SSRI) medications (fluoxetine, sertraline, escitalopram)
  Other Names: SSRI plus CBT; COMB
  Arms: Combination therapy (COMB)

SUMMARY:
Pediatric onset anxiety disorders (generalized anxiety, social anxiety, separation anxiety) are highly prevalent, and if untreated, are impairing into adolescence and adulthood. In the largest comparative efficacy study remission occurred in about 65% of children and adolescents treated with a combination of a selective serotonin reuptake inhibitors (SSRI) and cognitive behavioral therapy (CBT). In contrast, CBT without an SSRI achieved remission in 35% of children at 3 months and 45% at 6 months-a 30% and 20% difference, respectively. Despite the difference in remission rates, CBT alone is the preferred treatment of most patients and families. Lack of awareness of the significant difference in remission rates and concerns about medication side effects may drive patient and family preference even though SSRIs have a positive safety profile.

Critiques of CBT in the above study suggest that CBT was not as effective as it could be due to short treatment duration, restricted family involvement and limited exposure sessions. Would the combination of CBT and an SSRI still be superior to CBT only, if CBT was of longer duration, and included more family involvement and exposure sessions?

In the Partners in Care for Anxious Youth (PCAY) study, children and adolescents with an anxiety disorder ages 7-17 years followed in pediatric primary care clinics affiliated with three institution: Lurie Children's Hospital of Chicago, University of California Los Angeles and University of Cincinnati will be randomized to one of two treatment arms; either CBT only or CBT combined with an SSRI (either fluoxetine, sertraline, or escitalopram). CBT in PCAY will be 6 months in duration and include more family involvement, and more exposure opportunities than past trials. The 6-month acute treatment phase will be followed by 6 months of followup. The primary outcome will be anxiety symptom remission and reduction in impairment over 6 and 12-months.

DETAILED DESCRIPTION:
Anxiety disorders begin during childhood and adolescents, are extremely common, but are often under-diagnosed and under-treated. If untreated, pediatric anxiety disorders can be chronic and impairing into adulthood. The good news is that evidence-based treatments can be highly effective in reducing symptoms, and for a good number of children and adolescents, treatment can reduce anxiety symptoms to a minimum with marked improvement in function. In the largest comparative efficacy study, remission (minimal or no symptoms of anxiety), occurred in about 65% of children and adolescents treated with a combination of a selective serotonin reuptake inhibitor (SSRI) and cognitive behavioral therapy (CBT). In contrast, CBT without an SSRI achieved remission in 35% of children at 3 months and 45% at 6 months-a 30% and 20% difference, respectively.

Nonetheless, CBT alone is the preferred treatment of most patients and families. Lack of awareness of the significant difference in remission rates and concerns about medication side effects may drive patient and family preference, even though SSRIs have a positive safety profile.

In the study described above, CBT was limited in ways that might account for why it was less effective. CBT was shorter in duration, had fewer sessions, and less exposure opportunities than it was originally designed to have and had less family involvement than more current approaches. Given that patients and families prefer CBT, it is important to know if combination of CBT and an SSRI is truly superior to CBT only or whether fully implemented CBT can close the gap in remission rates with the combination of CBT and an SSRI. The study will also provide information about which children and adolescents achieve remission with CBT or CBT and an SSRI.

The Partners in Caring for Anxious Youth (PCAY) study will screen children and adolescents ages 7-17 years in pediatric primary care clinics affiliated with three institution: Lurie Children's Hospital of Chicago, University of California Los Angeles and University of Cincinnati. If a child screens positive with symptoms of an anxiety disorder, the patient and family will be offered an opportunity to learn about PCAY. If the family is interested in PCAY, a study staff person will provide information and answer any questions. If the patient and family want to enroll they will sign a consent form, complete an evaluation, and if eligible and willing to move forward, be randomized to either CBT or CBT plus an SSRI. The study team will work with the patient and family to connect to a therapist in the community to start CBT and if medication is part of treatment, work with the patient's pediatrician to begin medication. CBT will include up to 20 session of therapy and medication treatment will be a selective serotonin reuptake inhibitor (either fluoxetine, sertraline or escitalopram). The goal of treatment is for the child or adolescent with an anxiety disorder to reach remission and have a marked improvement in functioning. The first part of treatment lasts 6 months and there is then ongoing follow-up for an additional 6 months (12 months total). When the study is finished, the investigators hope to know if CBT and an SSRI is really superior to fully implemented CBT or not. The results of this study will inform patients, families, providers, payors and policy makers on the value of medication when combined with CBT.

ELIGIBILITY:
Inclusion Criteria

1. Ages 7-17 years (inclusive at time of consent/assent)
2. Primary Diagnostic and Statistical Manual, 5th Edition (DSM-5) diagnosis of separation anxiety disorder (SAD), and/or generalized anxiety disorder (GAD), and/or social anxiety disorder (SocAD) as determined by self-reported structured interview (MINI-KID) and confirmation by a study clinician.
3. Stable/treated Attention Deficit Hyperactivity Disorder (ADHD), combined or hyperactive impulsive subtypes
4. An available primary caretaker with ongoing patient contact who is legally able to provide consent
5. Medically cleared by a pediatric clinician including a negative urine pregnancy test for females of child-bearing age. Furthermore, female patients must agree to abstain from sexual activity or to use a reliable method of birth control as determined by pediatric clinician during the study.

Exclusion Criteria:

1. Patients with the following lifetime psychiatric disorders: moderate to severe autism, bipolar disorder, schizophrenia, or schizoaffective disorder, history of intellectual disability
2. Primary Attention Deficit Hyperactivity Disorder (ADHD), combined or hyperactive impulsive subtypes
3. Major depressive disorder with greater severity than anxiety disorder requiring treatment not provided in PCAY
4. Obsessive Compulsive Disorder (OCD) only (no co-occurring SAD, SocAD or GAD)
5. Patients with a major medical illness that would interfere with participation in the study (e.g., complex, and evolving medical treatments, or require frequent hospitalizations).
6. Patients who are pregnant as indicated by a positive pregnancy test or are sexually active and not using effective birth control.
7. Patients who pose a significant and imminent risk to self or to others.
8. Patients who experienced minimal or no change an adequate dose of evidenced-based medication treatment or CBT for their anxiety disorder.

   (See medication and CBT exclusions below)
9. Patients or caregiver(s) who do not speak English or Spanish. All materials and treatments will be available in Spanish and English.
10. Children and adolescents with complex psychiatric needs that cannot be managed in primary care and community settings as determined by study local Principal Investigator (PI) and provider teams.

Medication Exclusions

Fluoxetine

* 20 mg for at least 6 of 10 weeks in children <12 year
* 40 mg for at least 6 of 10 weeks in adolescents >12 years

Sertraline

* 100 for at least 6 of 10 weeks in children <12 years
* 150 for at least 6 of 10 weeks in adolescents >12 years

Citalopram

* 20 mg for at least 6 of 10 weeks in children >12 years
* 30 mg for at least 6 of 10 weeks adolescent > 12 years

Escitalopram

* 10 mg for at least 6 of 10 weeks in children <12 years
* 20 mg for at least 6 of 10 weeks in adolescent >12 years

Fluvoxamine

* 150 mg for at least 6 of 10 weeks in children <12 years
* 200 mg for at least 6 of 10 weeks in children < 12 year

CBT Exclusions

Failed a previous trial of verified CBT for anxiety disorders within the previous year judged adequate by ≥12 exposure-based CBT sessions

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 468 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression-Severity Scale (CGI-S) | The primary outcome is anxiety disorder remission based on a parent- and child-reported CGI-S rating of 1 (not at all ill) or 2 (borderline ill) at 6 months from first treatment visit
  The CGI-S score provides a global rating of anxiety symptom severity ranging from 1 (not at all ill) to 7 (extremely ill). The CGI-S is commonly used in clinical trials and will allow us to benchmark across prior studies in the field.
Child Anxiety Impairment Scale-Revised (CAIS-R) | Change in CAIS-R rating of anxiety-related impairment from baseline to 6 months post treatment
  The CAIS-R is a 47-item parent- and child-reported rating of the degree to which anxiety symptoms are impairing the child or adolescent's functioning. Scores range from 0-141 with higher scores indicate poorer functioning.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity Scale (CGI-S) | The primary outcome is anxiety disorder remission based on a parent- and child-reported CGI-S rating of 1 (not at all ill) or 2 (borderline ill) at 12 months from first treatment visit
  The CGI-S score provides a global rating of anxiety symptom severity ranging from 1 (not at all ill) to 7 (extremely ill). The CGI-S is commonly used in clinical trials and will allow us to benchmark across prior studies in the field.
Child Anxiety Impairment Scale-Revised (CAIS-R) | Change in CAIS-R rating of anxiety related impairment from baseline to 12 months post treatment
  The CAIS-R is a 47-item parent- and child-reported rating of the degree to which anxiety symptoms are impairing the child or adolescent's functioning. Scores range from 0-141 with higher scores indicate poorer functioning.

CONTACTS AND LOCATIONS:
Overall Officials: John Walkup, MD, Principal Investigator — Chair, Pritzker Department of Psychiatry and Behavioral Health
Locations (3):
- United States (3):
  - UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California
  - Lurie Children's Hospital and Affiliated Pediatric Practices, Chicago, Illinois
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
The final cleaned and locked data set that contains all the data used in conducting the analyses reported in the in the Patient Centered Outcome Research Institute (PCORI) Final Research Report and is fully de-identified in accordance with the the HIPAA Rule. These data include all baseline demographic and diagnostic data, baseline anxiety measures and repeated anxiety measures across the acute phase of the study. The data set will allow for replicating the primary outcomes and baseline moderators of the study's primary outcome. The data will be deposited in a PCORI designated repository within 3 years after the study has been completed and after acceptance by PCORI of the Final Research Report or publication of the key outcome paper(s) in a peer reviewed journal - whichever comes first.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be deposited in a PCORI designated repository within 3 years after the study has been completed and after acceptance of the by PCORI of the Final Research Report or publication of the key outcome paper(s) in a peer reviewed journal - which ever comes first.
Access Criteria: Individual investigators or teams of investigators seeking access to data from PCORI-funded studies must complete and submit a data request form to a PCORI-designated repository. The repository will independently review requests for data based on qualifications of the data requestors and the scientific merit of the request

REFERENCES:
- [Result] Walkup JT, Albano AM, Piacentini J, Birmaher B, Compton SN, Sherrill JT, Ginsburg GS, Rynn MA, McCracken J, Waslick B, Iyengar S, March JS, Kendall PC. Cognitive behavioral therapy, sertraline, or a combination in childhood anxiety. N Engl J Med. 2008 Dec 25;359(26):2753-66. doi: 10.1056/NEJMoa0804633. Epub 2008 Oct 30. PMID 18974308
- [Result] Piacentini J, Bennett S, Compton SN, Kendall PC, Birmaher B, Albano AM, March J, Sherrill J, Sakolsky D, Ginsburg G, Rynn M, Bergman RL, Gosch E, Waslick B, Iyengar S, McCracken J, Walkup J. 24- and 36-week outcomes for the Child/Adolescent Anxiety Multimodal Study (CAMS). J Am Acad Child Adolesc Psychiatry. 2014 Mar;53(3):297-310. doi: 10.1016/j.jaac.2013.11.010. Epub 2013 Nov 28. PMID 24565357
- [Result] Peris TS, Compton SN, Kendall PC, Birmaher B, Sherrill J, March J, Gosch E, Ginsburg G, Rynn M, McCracken JT, Keeton CP, Sakolsky D, Suveg C, Aschenbrand S, Almirall D, Iyengar S, Walkup JT, Albano AM, Piacentini J. Trajectories of change in youth anxiety during cognitive-behavior therapy. J Consult Clin Psychol. 2015 Apr;83(2):239-52. doi: 10.1037/a0038402. Epub 2014 Dec 8. PMID 25486372
- [Result] Strawn JR, Dobson ET, Mills JA, Cornwall GJ, Sakolsky D, Birmaher B, Compton SN, Piacentini J, McCracken JT, Ginsburg GS, Kendall PC, Walkup JT, Albano AM, Rynn MA. Placebo Response in Pediatric Anxiety Disorders: Results from the Child/Adolescent Anxiety Multimodal Study. J Child Adolesc Psychopharmacol. 2017 Aug;27(6):501-508. doi: 10.1089/cap.2016.0198. Epub 2017 Apr 6. PMID 28384010
- [Result] Rynn MA, Walkup JT, Compton SN, Sakolsky DJ, Sherrill JT, Shen S, Kendall PC, McCracken J, Albano AM, Piacentini J, Riddle MA, Keeton C, Waslick B, Chrisman A, Iyengar S, March JS, Birmaher B. Child/Adolescent anxiety multimodal study: evaluating safety. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):180-90. doi: 10.1016/j.jaac.2014.12.015. Epub 2014 Dec 31. PMID 25721183